CLINICAL TRIAL: NCT06789614
Title: Comparison of the Effect of Cyclizine Versus Metoclopramide on Gastric Residual Volume in Patients Undergoing Bariatric Surgery: A Randomized Double-blinded Clinical Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatema alzhraa Mohammed mohammadeen, Doctor, Cairo University
Other Study IDs: GRS in bariatric surgery
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery
Keywords: GRV, Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cyclizine group: will receive intravenous Cyclizine (50 mg) in a 10 mL syringe.
  Interventions: Drug: intravenous CYCLIZINE ,Metaclopromide
- Metoclopramide group: participants will receive intravenous Metoclopramide (10 mg) in a (10 mL )syringe.

INTERVENTIONS:
Drug: intravenous CYCLIZINE ,Metaclopromide — US giuded measure of GRV in bariatrics surgery upon recieving drugs of study
  Groups: Cyclizine group

SUMMARY:
The aim of this work is to compare the effects metoclopramide versus Cyclizine withing the context of multimodal antiemetic strategy on GRV in patients scheduled for bariatric surgery.

DETAILED DESCRIPTION:
Patients undergoing bariatric surgery report significant postoperative nausea and vomiting (PONV), which contributes to delayed oral intake and mobilization with a subsequent prolonged hospital length of stay. (1) The high incidence of PONV after bariatric surgery is referred to several factors such as obesity, prevalence of hiatal hernia, direct gastric irritation by surgical trauma, blood, and secretions, abdominal insufflation, increased surgical duration of > 1 hour, and the use of opioids. (2,3) The latest consensus guidelines for prophylaxis against PONV recommended the use of > 2 prophylactic drugs in patients with > 2 risk factors for PONV (4). A considerable proportion of patients undergoing bariatric surgery have > 2 risk factors (laparoscopic bariatric procedure - young age - non-smokers - opioid use). The first and second lines for prophylaxis are commonly 5HT-3 antagonist (e.g., ondansetron) and dexamethasone. However, there is no clear evidence for the superiority of either of the 3rd line drugs over the other. Several groups of drugs are suggested as 3rd line drugs such as dopamine receptor antagonists (e.g., metoclopramide) (5) ; histamine antagonists (e.g., prochlorperazine and Cyclizine) (6) , anticholinergics (such as scopolamine) (7) and neurokinin antagonists (such as Fosaprepitant) (8) .

Metoclopramide acts centrally by blocking dopamine receptors in the CTZ and vomiting centre and peripherally by shortening bowel transit time and in high doses blocks serotonin receptors. (9) Cyclizine is a piperazine derivative. It is an antihistamine i.e (H1)- receptor antagonist, and also has some effect on the dopamine (D2) and cholinergic receptors and inhibits integrative function of the vestibular nuclei. (10,11) measurement of the Gastric residual volume (GRV) has been widely used in perioperative medicine the last few years especially with the increased interest in point-of-care ultrasound. GRV is a predictor of PONV (12). Furthermore, several reports used GRV as an index of the prokinetic efficiency of antiemetic drugs (13,14) The aim of this study is to evaluate the effects of metoclopramide versus Cyclizine, within the context of multimodal antiemetic strategy, on GRV in patients scheduled for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria

* ● Age (18 - 40).

  * Body mass index (BMI) 40 to 50 kg/m2.4
  * American Society of Anaesthesiologist (ASA) - physical status III.
  * Patients undergoing bariatric surgery.
  * Non smokers.

Exclusion Criteria:

* ● Refusal of the patient

  * Deviation from fasting times
  * Patients with empty stomach
  * Body mass index (BMI) less than 40s kg/m2
  * American Society of Anesthesiologists (ASA) physical status class IV.
  * Systemic diseases may cause delayed gastric emptying (eg: myopathies and myasthenia gravis).
  * Patients with gastrointestinal diseases which impact the gastric emptying such as hiatus hernia, intestinal disease and gastro-oesophageal reflux disease and patients with history of upper gastrointestinal surgeries.
  * Use of other medications known to affect gastric motility or secretions (Diphenoxylate, Atropine& Imodium) or secretions.
  * Allergy to macrolide or metoclopramide. • a considerable proportion of patients with obesity have diabetes and thus, they cannot be excluded from the study. However, we would exclude patients with long standing diabetes (more than 5 years) who are likely to have delayed gastric emptying. Furthermore, this is a randomized controlled trial and the randomization usually overcomes these points and the demographic data would be displayed in the results to clarify whether there is a balance between the two groups or not.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: morbidely obese ASA2-3
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Estimated Gastric volume (mL) | 1 hour after administration of the study drugs
  Estimated Gastric volume (mL) based on the antral CSA in the RLD (CSARLD) by gastric ultrasonic 1 hour after administration of the study drugs.

SECONDARY OUTCOMES:
● Incidence of PONV | 24 hours
  ● Incidence of PONV in the 1st postoperative 24 hours (who receive the rescue antiemetic when the PONV grade reaches ≥ 2 or the 10_points Likert score reaches ≥ 4).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 1. Celio A, Bayouth L, Burruss MB, Spaniolas K. Prospective assessment of postoperative nausea early after bariatric surgery. Obes Surg. 2019 Mar; 29(3):858- 861. — https://link.springer.com/article/10.1007/s11695-018-3605-1
- See also: Naeem Z, Chen IL, Pryor AD, Docimo S, Gan TJ, Spaniolas K. Antiemetic prophylaxis and anesthetic approaches to reduce postoperative nausea and vomiting in bariatric surgery patients: a systematic review. Obesity surgery. 2020 Aug;30:3188-200. — https://link.springer.com/article/10.1007/s11695-020-04683-1
- See also: 4. Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC. Fourth consensus guidelines for the management of postoperative nausea and vomiting. Anesthesia & Analgesia. — https://journals.lww.com/anesthesia-analgesia/fulltext/2020/08000/Fourth_Consensus_Guidelines_for_the_Management_of.16.aspx?context=FeaturedArticles&collectionId=6